CLINICAL TRIAL: NCT07396636
Title: Machine Learning-Assisted Intraoperative Hypotension Management: Developing Personalized Treatment Recommendations
Brief Title: Machine Learning-Assisted Management of Intraoperative Hypotension for Personalized Treatment
Acronym: HYPOGUARD
Status: Not yet recruiting | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, MD, Associate Professor, Nevsehir Public Hospital
Other Study IDs: E2-25-12078
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intraoperative Hypotension; Perioperative Care; Hemodynamic Monitoring; Blood Pressure; Anesthesia, General
Keywords: Intraoperative hypotension; Machine learning; Personalized treatment; Clinical decision support; Hemodynamic instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraoperative hypotension, defined as a drop in blood pressure during surgery, is a frequent event in patients undergoing general anesthesia. Even brief episodes of low blood pressure may reduce blood flow to vital organs such as the brain, heart, and kidneys, and have been associated with an increased risk of postoperative complications, prolonged recovery, and worse clinical outcomes. Despite its clinical importance, the management of intraoperative hypotension is often based on general guidelines and individual clinician experience rather than patient-specific physiological mechanisms.

Low blood pressure during surgery can occur for different underlying reasons, including reduced circulating blood volume, excessive vasodilation caused by anesthetic agents, impaired heart contractility, or abnormalities in heart rate. In routine practice, these mechanisms are not always clearly distinguished, and similar treatment strategies may be applied to patients with different physiological causes of hypotension. As a result, the response to treatment can vary widely between patients.

This prospective observational study aims to improve the understanding of intraoperative hypotension by collecting detailed hemodynamic data during surgery and analyzing these data using machine learning methods. The study is designed to observe current clinical practice without altering or interfering with routine patient care. All decisions regarding anesthesia management and treatment of hypotension will be made by the attending anesthesiologists according to standard clinical practice. The research team will not provide treatment recommendations during surgery.

Adult patients undergoing elective surgery under general anesthesia with continuous invasive arterial blood pressure monitoring will be included. During the intraoperative period, blood pressure, heart rate, cardiac output, stroke volume, systemic vascular resistance, and other advanced hemodynamic parameters will be continuously recorded at regular intervals. When hypotension occurs, the onset, duration, and severity of the episode will be documented, along with the treatment applied, such as fluid administration, vasopressor agents, or inotropic medications. The time required for blood pressure to recover to an acceptable level will also be recorded.

The collected data will be analyzed using machine learning techniques to identify distinct subtypes of intraoperative hypotension based on physiological patterns. These subtypes may reflect different underlying mechanisms, such as hypovolemia, vasodilation, myocardial depression, or heart rate-related causes. In addition, the study will evaluate how different treatment strategies perform across these hypotension subtypes and how quickly hemodynamic stability is restored.

Patient-related factors such as age, sex, body mass index, physical status classification, and comorbid conditions will also be examined to determine their relationship with the occurrence, severity, and treatment response of hypotension episodes. By combining patient characteristics, physiological data, and treatment responses, the study aims to generate data-driven insights into personalized hypotension management.

The ultimate goal of this research is to support the development of individualized treatment recommendations for intraoperative hypotension based on objective physiological data rather than a one-size-fits-all approach. The findings of this study are expected to provide a strong scientific foundation for future clinical decision-support systems that can assist anesthesiologists in selecting the most appropriate treatment strategy for each patient. By improving the precision of blood pressure management during surgery, this approach has the potential to enhance patient safety and perioperative outcomes while maintaining standard clinical workflows.

DETAILED DESCRIPTION:
Intraoperative hypotension, commonly defined as a decrease in arterial blood pressure during surgery, is a frequent and clinically important event in patients undergoing general anesthesia. Numerous studies have shown that even brief periods of low blood pressure may be associated with impaired organ perfusion and an increased risk of postoperative complications, including acute kidney injury, myocardial injury, stroke, prolonged hospital stay, and increased mortality. Despite growing awareness of its clinical impact, the optimal management of intraoperative hypotension remains an ongoing challenge in anesthetic practice.

Current approaches to intraoperative blood pressure management are largely based on general thresholds, guideline recommendations, and the individual experience of anesthesiologists. In routine clinical practice, hypotension is often treated with fluid administration, vasopressor agents, inotropic drugs, or combinations of these interventions. However, hypotension is not a single, uniform clinical entity. It may arise from different underlying physiological mechanisms, such as hypovolemia, anesthetic-induced vasodilation, myocardial depression, or heart rate abnormalities. These mechanisms may coexist or change dynamically during surgery, making clinical decision-making complex.

In many cases, similar treatment strategies are applied to patients with different physiological causes of hypotension, which may lead to variable treatment responses. For example, fluid administration may be effective in patients with hypovolemia but less beneficial or even harmful in patients with predominant vasodilation or impaired cardiac function. Likewise, vasopressor therapy may rapidly restore blood pressure in vasodilatory hypotension but may not adequately address hypotension caused by low cardiac output. This highlights the need for a more individualized, physiology-based approach to intraoperative hypotension management.

Recent advances in perioperative monitoring have enabled continuous, high-resolution recording of arterial blood pressure and advanced hemodynamic parameters, such as cardiac output, stroke volume, and systemic vascular resistance. At the same time, developments in machine learning and artificial intelligence have created new opportunities to analyze large and complex datasets, identify hidden patterns, and generate data-driven insights that may not be apparent through traditional statistical methods.

The primary aim of this prospective observational study is to improve the understanding of intraoperative hypotension by integrating detailed hemodynamic monitoring with machine learning-based analysis. Rather than focusing on a single blood pressure threshold or isolated variables, this study seeks to characterize hypotension episodes as dynamic physiological events and to identify distinct hypotension subtypes based on underlying hemodynamic patterns.

This study is designed as a non-interventional, observational investigation and does not alter routine clinical care. All anesthesia management decisions, including the prevention and treatment of hypotension, will be made by the attending anesthesiologists according to standard clinical practice and institutional protocols. The research team will not provide real-time recommendations or influence clinical decision-making during surgery. The role of the research team is limited to systematic data collection, data processing, and post hoc analysis.

Adult patients (≥18 years of age) undergoing elective surgical procedures under general anesthesia will be included. Continuous invasive arterial blood pressure monitoring is required for inclusion, as it allows precise, beat-to-beat assessment of blood pressure and waveform-derived hemodynamic variables. Emergency surgeries, patients with severe circulatory shock, advanced cardiac dysfunction, or conditions that prevent reliable hemodynamic measurements will be excluded to ensure data quality and patient safety.

During the intraoperative period, arterial blood pressure, heart rate, cardiac output, cardiac index, stroke volume, stroke volume index, systemic vascular resistance, and related dynamic preload variables will be continuously recorded at predefined time intervals. Hypotension will be defined as a mean arterial pressure below a clinically relevant threshold sustained for a minimum duration. When hypotension occurs, the onset time, duration, severity, and frequency of each episode will be documented.

In addition to physiological data, detailed information regarding therapeutic interventions will be collected. This includes the type and amount of intravenous fluids administered, the use of vasopressor agents or inotropic drugs, dosing strategies, and the timing of interventions relative to hypotension onset. The response to treatment will be assessed by measuring the time required for blood pressure to return to predefined target values and by evaluating changes in other hemodynamic parameters following intervention.

Machine learning techniques will be applied to the collected dataset to identify patterns and clusters within hypotension episodes. Unsupervised learning methods, such as clustering algorithms, will be used to classify hypotension events into subtypes based on hemodynamic profiles. These subtypes are expected to reflect different dominant physiological mechanisms, such as volume depletion, vasodilation, myocardial depression, or heart rate-related hypotension.

In parallel, supervised learning models will be used to explore relationships between patient characteristics, hemodynamic patterns, treatment strategies, and treatment responses. Variables such as age, sex, body mass index, physical status classification, comorbidities, and surgical characteristics will be analyzed to determine their association with hypotension occurrence, subtype distribution, and responsiveness to specific interventions.

One of the key objectives of this study is to evaluate whether certain treatments are more effective for specific hypotension subtypes or patient profiles. By analyzing treatment response times and hemodynamic recovery patterns, the study aims to generate evidence supporting more targeted and individualized treatment strategies. These analyses will not be used to guide patient care during the study but will form the basis for future hypothesis generation and interventional research.

All collected data will be anonymized and stored securely in accordance with data protection regulations. Only authorized members of the research team will have access to the dataset. The study will adhere to ethical principles for clinical research, and informed consent will be obtained from all participants prior to inclusion.

The ultimate goal of this research is to contribute to the development of data-driven, personalized approaches to intraoperative blood pressure management. By combining high-quality physiological data with advanced analytical methods, this study aims to provide a deeper understanding of intraoperative hypotension and its heterogeneous nature. In the long term, the findings may support the development of clinical decision-support systems that assist anesthesiologists in selecting the most appropriate treatment strategy for each patient based on real-time physiological information.

Such systems have the potential to improve patient safety, reduce the burden of postoperative complications, and enhance the quality of perioperative care without replacing clinical judgment. Instead, they are intended to complement the expertise of anesthesiologists by providing objective, individualized insights derived from complex data patterns. This study represents an important step toward more precise, personalized, and physiology-guided management of intraoperative hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Patients scheduled for elective surgical procedures
* Procedures performed under general anesthesia
* Availability of continuous invasive arterial blood pressure monitoring during the intraoperative period
* Planned surgical duration of at least 2 hours
* Ability to provide written informed consent for participation in the study

Exclusion Criteria:

* Emergency surgery
* Diagnosis of sepsis, septic shock, or advanced cardiogenic shock
* Cardiac rhythm disturbances that prevent reliable hemodynamic measurements (e.g., atrial fibrillation)
* Severe left ventricular dysfunction or advanced heart failure (ejection fraction <30%)
* Inability to maintain intraoperative arterial cannulation due to technical or clinical reasons
* Inability to provide informed consent (e.g., cognitive impairment or refusal to participate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from adult patients undergoing elective surgical procedures under general anesthesia at a tertiary care hospital. Participants will be selected from operating rooms where continuous invasive arterial blood pressure monitoring is routinely used as part of standard anesthetic care. The study will include patients managed according to usual clinical practice by attending anesthesiologists, without any protocol-driven intervention. Data will be collected prospectively during the intraoperative period from routine monitoring systems and anesthesia records. The population reflects a real-world perioperative setting in which intraoperative hypotension is commonly encountered and managed using standard hemodynamic monitoring and treatment strategies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hypotension endotype classification (hemodynamic subtype) per hypotension episode | Intraoperative period (from anesthesia induction to the end of surgery)
  For each intraoperative hypotension episode (defined as mean arterial pressure [MAP] <65 mmHg lasting ≥1 minute, or a ≥30% decrease from baseline), the episode will be assigned to a hemodynamic endotype based on invasive arterial waveform-derived parameters recorded using MostCare® (Vygon, France), including MAP, SAP, DAP, HR, CO, CI, SV, SVI, SVR, SVRI, SVV, PPV, and SPV, sampled every 30 seconds.
  The outcome is the endotype label assigned to each episode, reported as a categorical classification with the following levels:
  Hypovolemic endotype, Vasodilatory endotype, Myocardial depression endotype and Bradycardic endotype.

SECONDARY OUTCOMES:
Time to hemodynamic stabilization after treatment of intraoperative hypotension | Intraoperative period (from anesthesia induction to the end of surgery)
  For each intraoperative hypotension episode (mean arterial pressure [MAP] <65 mmHg lasting ≥1 minute), the time interval from initiation of therapeutic intervention (fluid administration, vasopressor, or inotropic therapy) to achievement of MAP ≥65 mmHg will be recorded.
  Hemodynamic data will be obtained from invasive arterial blood pressure monitoring using MostCare® (Vygon, France), with parameters sampled every 30 seconds. The timestamp of treatment initiation will be matched with arterial pressure recordings to calculate recovery time.
Correlation between patient characteristics and intraoperative hypotension burden | Intraoperative period (from anesthesia induction to the end of surgery)
  Correlation between patient characteristics (age, sex, BMI, ASA class, comorbidities, chronic antihypertensive use) and intraoperative hypotension burden (number of hypotension episodes per patient, total duration of hypotension in minutes, and minimum MAP during surgery)
  Age (years), sex (male/female), BMI (kg/m²), ASA class (I-IV), comorbidities (presence/absence of hypertension, diabetes, CAD, etc.), chronic antihypertensive medication use (yes/no); collected from the anesthesia record and hospital electronic medical record.
  Number of intraoperative hypotension episodes per patient (count), total duration of hypotension per patient (minutes), minimum intraoperative MAP (mmHg); derived from continuous invasive arterial pressure monitoring using MostCare® (Vygon, France), sampled every 30 seconds.
Performance of AI-based personalized hypotension treatment recommendation model | Intraoperative period (from anesthesia induction to the end of surgery)
  Performance of machine learning models (Decision Tree, Random Forest, XGBoost) in predicting the most effective treatment strategy (fluid, vasopressor, inotrope, or combination) for intraoperative hypotension episodes, based on patient characteristics and hemodynamic endotype, compared to observed real-world treatment response (time to MAP ≥65 mmHg and hemodynamic stabilization).
  Patient characteristics: age (years), sex, BMI (kg/m²), ASA class, comorbidities, chronic antihypertensive use (yes/no), collected from anesthesia record/EMR.
  Hemodynamic endotype per hypotension episode, derived from invasive arterial waveform monitoring with MostCare® (Vygon, France), using MAP, SAP, DAP, HR, CO, CI, SV, SVI, SVR, SVRI, SVV, PPV, SPV sampled every 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Yazar, MD, PhD, Assoc. Prof, Study Director — Konya City Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers due to the nature of high-resolution intraoperative hemodynamic data and institutional data governance policies. All analyses will be conducted on anonymized datasets within the research team, and only aggregate results will be reported.